CLINICAL TRIAL: NCT06708741
Title: Regime for Vitamin D Maintenance in Post-Operative Patients (D-ECISIVE) Randomized Controlled Trial
Brief Title: Regime for Vitamin D Maintenance in Post-Operative Patients
Acronym: D-ECISIVE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sengkang General Hospital (Other)
Collaborators: Hyphens Pharma Pte Ltd (Industry)
Responsible Party: Principal Investigator, Koh Hong Xiang Frederick, Consultant Colorectal Surgeon, Sengkang General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024-3998
Record Dates: First submitted 2024-10-21; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D supplementation (Experimental): High dose oral vitamin D supplementation (50,000 IU/once a month)
  Interventions: Drug: Vitamin D
- Standard-of-care Arm (No Intervention): standard of care arm where vitamin D levels are not actively acted upon

INTERVENTIONS:
Drug: Vitamin D — High dose oral vitamin D supplementation (50,000 IU/once per month)
  Other Names: D-cure
  Arms: Vitamin D supplementation

SUMMARY:
Vitamin D plays a significant part calcium and phosphate haemostasis, thus, intrinsically critical for bone health. Increasing evidence also reveal that insufficient serum vitamin D levels also result in poor muscle health with such individuals having a compromised muscle building potential (4 times slower muscle building).

Muscle health is a critical component of a post-surgical patient recovery, with impaired muscle function leading to reduced functional ability, resulting in a poorer quality of life. Poor muscle health also has negative repercussion on survivability, with reduced overall, and disease-specific survival, especially shown in cancer patients. Thus, maintenance of vitamin D levels post-surgery may be more critical than previously thought.

DETAILED DESCRIPTION:
This study is performed in Singapore (outside the US) and the medication, while it is a FDA approved medication, is not manufactured in the US for the trial purpose and the indications of use in this trial is not new.

The investigators would be recruiting patients aged 21-65 years who have undergone major surgery (defined by the NICE criteria) and who are able to provide informed consent, accept to take vitamin D supplements post-operatively and have their serum vitamin D levels checked periodically.

The investigators will excluded patients who have undergone minor procedures (Table code <4a), those who have a history of chronic kidney disease/end staged renal failure, known hyperparathyroidism, are non-ambulatory independently and have had known allergies to the commercially available high dose vitamin D formulations.

High dose oral vitamin D supplementation (50,000 IU/week for 8 weeks) is the current recommended dose for individuals with vitamin D insufficiency of deficiency and is currently being used for some prehabilitation programmes due to the quick repletion of vitamin D levels to improve muscle gain during the short prehabilitation window prior to surgery.

Using the same dose once a month would provide a significantly less vitamin D supplementation, especially with individuals who have had their vitamin D levels repleted in the preoperative phase. This will be compared against a control who are randomised to standard-of-care (SOC) where high dose vitamin D maintenance is not prescribed.

The unmet clinical need is the still unknown, unstandardised vitamin D supplementation regime. There are current no clinical consensus on vitamin D supplementation after patients who have undergone major surgery.

ELIGIBILITY:
Inclusion Criteria:

* Serum 25-hydroxyvitamin D levels between 30-50ng/ml at 4-6 weeks after operation
* aged 21-65 years
* ability to provide informed consent
* accepts to take vitamin D supplements post-operatively and
* have their serum vitamin D levels checked periodically.

Exclusion Criteria:

* They have undergone minor procedures (Table code <4a)
* have a history of chronic kidney disease/end staged renal failure
* have previous history of ureteric/kidney stones
* known hyperparathyroidism
* are non-ambulatory independently
* have had known allergies to the commercially available high dose vitamin D formulations.
* Vulnerable personnel would be excluded from the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
serum 25-hydroxyvitamin D levels at 3-months post-intervention | 3 months after initiation
  serum 25-hydroxyvitamin D levels at 3-months post-intervention

SECONDARY OUTCOMES:
serum 25-hydroxyvitamin D levels compared to SOC at 6-months post-intervention. | 6 months after initiation
  serum 25-hydroxyvitamin D levels compared to SOC at 6-months post-intervention.
serum 25-hydroxyvitamin D levels compared to SOC at 12-months post-intervention. | 12 months after initiation
  serum 25-hydroxyvitamin D levels compared to SOC at 12-months post-intervention.
functional outcome measures at 3-months post-intervention | 3-months after intiation
  functional outcome measures at 3-months post-intervention
functional outcome measures at 6-months post-intervention | 6 months after initiation
  functional outcome measures at 6-months post-intervention
functional outcome measures at 12-months post-intervention | 12 months after initiation
  functional outcome measures at 12-months post-intervention
muscle quality (Ultrasound+MuscleSound™ evaluation) at 3-months post-intervention | 3 months after intiation
  muscle quality (Ultrasound+MuscleSound™ evaluation) at 3-months post-intervention
muscle quality (Ultrasound+MuscleSound™ evaluation) at 6-months post-intervention | 6 months after initiation
  muscle quality (Ultrasound+MuscleSound™ evaluation) at 6-months post-intervention
muscle quality (Ultrasound+MuscleSound™ evaluation) at 12-months post-intervention | 12 months after initiation
  muscle quality (Ultrasound+MuscleSound™ evaluation) at 12-months post-intervention
quality of life (EQ5D-3L) at 3-months post-intervention | 3 months after intiation
  quality of life (EQ5D-3L) at 3-months post-intervention
quality of life (EQ5D-3L) at 6-months post-intervention | 6 months after initiation
  quality of life (EQ5D-3L) at 6-months post-intervention
quality of life (EQ5D-3L) at 12-months post-intervention | 12 months after initiation
  quality of life (EQ5D-3L) at 12-months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Frederick H Koh, FRCS, PhD, Principal Investigator — Sengkang General Hospital
Locations (1):
- Sengkang General Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
only centrally available to the PI